CLINICAL TRIAL: NCT04427319
Title: A Randomised Double-blind Clinical Trial to Analyse the Efficacy of Short-term β-Alanine Supplementation in Performance Outcomes of Road Professional Endurance Cyclists
Brief Title: The Efficacy β-Alanine Supplementation in Performance Outcomes of Road Professional Endurance Cyclists
Acronym: ELITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00014
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Supplementation; Cyclists
MeSH Terms: interventions — Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Product: β-Alanine Supplementation strategy: 5 g, four times a day with main meals, for 7 days after the initial evaluation and until the end of the study.
  Interventions: Dietary Supplement: β-alanine
- Placebo group (Placebo Comparator): Product: wheat semolina Supplementation strategy: 5 g, four times a day with main meals, for 7 days after the initial evaluation and until the end of the study.
  Interventions: Dietary Supplement: wheat semolina

INTERVENTIONS:
Dietary Supplement: β-alanine — 7 days of consumption
  Arms: Experimental group
Dietary Supplement: wheat semolina — 7 days of consumption
  Arms: Placebo group

SUMMARY:
A double-blind, placebo-controlled, randomised, with two arms (product and placebo) unicentric clinical trial to analyse the efficacy on physical performance parameters of a product designed for sport during a lapse of two weeks (7 days).

DETAILED DESCRIPTION:
After recruitment, subject will be randomised and allocated to one group of the 2 study arms: treatment group or control group (placebo).

A simple randomisation will be performed using software by a random number generator, and assigned to participants.

ELIGIBILITY:
Inclusion Criteria:

* Not respecting rest the day before physical tests.
* Not being in a fasted state (at least 2 h from last meal).
* Having consumed stimulants acutely before the trial, or under drug treatment affecting perceived effort of the trial.
* Not being available to perform every trial on the same conditions at the same time of the day.
* Not sticking to the same diet, 24 h before each trial.

Exclusion Criteria:

* Adverse event
* Protocol violation
* Lost to follow-up
* Allergy to any of the components of the treatment or placebo product. This includes allergy to β-alanine, wheat, soy, nuts (including peanuts), sesame and its byproducts.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | Change of baseline rate of perceived exertion at seven days
  Rate of perceived exertion

SECONDARY OUTCOMES:
Performance outcomes | It will be measured on two different occasions. Day one and seven days later.
  Physical performance is measured by direct variables: mean power output (MPO) and peak power output by ergometer (Cyclus 2) together with cadence.
Paresthesia test | It will be measured on three different occasions. Twice on day 1 (before and after consumption) and seven days after.
  Visual analogue scale (1-10)
Microcapillary blood | It will be measured on two different occasions. Day one and seven days later.
  This test provides biochemical variables (ABL90FLEX).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Pinero S, Ramos-Campo DJ, Lopez-Roman FJ, Ortolano R, Torregrosa-Garcia A, Luque-Rubia AJ, Ibanez-Soroa N, Andreu-Caravaca L, Avila-Gandia V. Effect of high-dose beta-Alanine supplementation on uphill cycling performance in World Tour cyclists: A randomised controlled trial. PLoS One. 2024 Sep 3;19(9):e0309404. doi: 10.1371/journal.pone.0309404. eCollection 2024. PMID 39226288